CLINICAL TRIAL: NCT04619381
Title: Investigation of the Causes of Health Disparities in African Americans With Coronary Artery Disease on Clopidogrel
Brief Title: Causes of Health Disparities in African Americans With Coronary Artery Disease on Clopidogrel
Status: Withdrawn | Type: Observational
Why Stopped: The study funding was dropped with no patients enrolled
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Aaron Aday, Instructor in Medicine Division of Cardiovascular Medicine, Vanderbilt University Medical Center
Other Study IDs: 171699
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: African American; Coronary Artery Disease; Anti Platelet
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African Americans with Coronary Artery Disease: African Americans with Coronary Artery Disease and currently taking clopidogrel
  Interventions: Behavioral: CORONARY ARTERY DISEASE AND CLOPIDOGREL: PATIENT SURVEY

INTERVENTIONS:
Behavioral: CORONARY ARTERY DISEASE AND CLOPIDOGREL: PATIENT SURVEY — Survey is a non-standardized assessment of demographics, medication compliance and reasons for non- compliance.

SUMMARY:
African Americans with coronary artery disease who have been prescribed clopidogrel (also known as Plavix), an antiplatelet drug will be enrolled. The purpose of this study is to help identify why African Americans are at an increased risk of having a major heart attack or stroke after a common procedure to open up blocked arteries with stents. The knowledge to be gained from this study includes:

1. A better understanding of the metabolism of the antiplatelet drug, clopidogrel, and abnormal platelet function in African Americans; this understanding may provide a basis for potential future therapy
2. A better understanding of challenges to taking clopidogrel as prescribed by a doctor and opinions about a genetic test related to this medicine.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Sex: Male and Female
3. Race: Self-identified as African American
4. History of percutaneous coronary intervention in the past 12 months
5. Currently taking aspirin and clopidogrel for at least one month and up to one year
6. English speaking

Exclusion Criteria:

1. Use of nonsteroidal anti-inflammatory drugs
2. Pregnancy will be excluded in women of child-bearing potential using urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant population will be recruited from routine care clinic/physician visits
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Participant Adherence to Plavix as Measured by Clopidogrel Metabolites in Plasma | baseline
  Participant adherence to Plavix as measured by clopidogrel metabolite in plasma by liquid chromatography-tandem mass spectrometry. Clopidogrel non-adherence will be defined as plasma concentration of inactive carboxyl metabolite <5,000 ng/mL.
Clopidogrel resistance | baseline
  Participant resistance to Plavix as measured by DNA analysis will be conducted to determine CYP2C19*2 loss of function (LOF) status. In addition, platelet function will be measured using the VerifyNow-P2Y12 point-of-care assay.
Platelet function | baseline
  Platelet function will be measured using the VerifyNow-P2Y12 point-of-care assay.
Patient-level barriers to implementation of routine pharmacogenomic testing for antiplatelet therapy | baseline
  Subjects will also complete a survey about clopidogrel adherence as well as their knowledge and attitudes about pharmacogenomic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Aday, MD, Principal Investigator — VUMC
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No